CLINICAL TRIAL: NCT03520751
Title: Phase I/IIa Trial Evaluating scAAV1.tMCK.NTF3 for Treatment of Charcot-Marie-Tooth Neuropathy Type 1A (CMT1A)
Brief Title: Phase I/IIa Trial of scAAV1.tMCK.NTF3 for Treatment of CMT1A
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Zarife Sahenk, Principal Investigator, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-01287
Record Dates: First submitted 2018-04-20; First posted 2018-05-11 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Charcot-Marie-Tooth Neuropathy Type 1A
Keywords: CMT1A; scAAV1.tMCK.NTF3; NTF3
MeSH Terms: conditions — Charcot-Marie-Tooth Disease | interventions — Disease Vectors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose (8.87e11 vg/kg) (Experimental): Three patients age 18-35 will receive intramuscular injection of recombinant AAV1 carrying a human NFT3 gene under the control of the tMCK promoter (scAAV1.tMCK.NTF3) distributed bilaterally between both limbs at a dose of 8.87e11 vg/kg.
  Interventions: Drug: scAAV1.tMCK.NTF3

INTERVENTIONS:
Drug: scAAV1.tMCK.NTF3 — gene vector
  Other Names: Neurotrophin Factor 3 (NTF3) vector

SUMMARY:
This clinical trial is an open-label one-time injection dose study in which scAAV1.tMCK.NTF3 will be administered by intramuscular injections into muscles in both legs in CMT1A subjects with PMP22 gene duplication. Three subjects ages 18 to 35 years receiving (8.87e11 vg/kg) will be enrolled.

DETAILED DESCRIPTION:
This clinical trial is an open-label, one-time injection study in which scAAV1.tMCK.NTF3 will be administered by intramuscular injections into the medial and lateral heads of gastrocnemius, tibialis anterior, and rectus femoris muscles in both legs in CMT1A subjects with PMP22 gene duplication. Three CMT1A patients, 18 to 35 years of age will be enrolled into one cohort in this trial. These adult subjects will be enrolled at an effective dose (8.87e11 vg/kg) based on a qPCR titer using linearized standards, equivalent to 4.00x1012 vg/kg based on a qPCR titer using supercoiled standards) distributed bilaterally between both limbs in Cohort 1. Post-gene transfer monitoring will include follow up visits on days 7, 14, 30, 60, 90, 120, and months 6, 9, 12, 15, 18 and 24 following gene transfer. Safety is the primary endpoint for this clinical gene transfer trial. Stopping criteria are based on development of unacceptable toxicity defined as the occurrence of any one Grade III or higher, unanticipated, treatment-related toxicity. The secondary endpoint is efficacy defined as halting of the decline in functional and sensory abilities measured by the CMT Pediatric Scale (CMTPedS) at 2 years post gene transfer. The CMTPedS is an 11-item scale comprised of the Functional Dexterity Test, Nine-Hole Peg Test (9HPT), hand grip, foot plantar flexion, foot dorsiflexion, pinprick sensation, vibration sensation, the Bruininks Oseretsky Test- Balance assessment, gait assessment, long jump, and six-minute walk test (6MWT). Exploratory outcome measures will include 10 meter run/walk timed test (10M), 100 meter timed test (100M), peroneal and ulnar CMAP amplitude and sensory and motor conduction velocities, a revised sensory testing to increase sensitivity for pinprick, touch-test and vibration assessments, visual analogue scales for pain and fatigue, Short Form Health Survey (SF-36) as Quality of Life measure, and circulating NT-3 levels.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18- 35 years old inclusive with CMT1A will be enrolled
* Must exhibit a 1.5 Mb duplication at 17p11.2 inclusive of the peripheral myelin protein 22 (PMP22) gene
* Males and females of any ethnic or racial group
* Must exhibit weakness of the ankle dorsiflexion muscle (but has full ROM against gravity and is able to stand on heels 3 seconds or greater)
* Abnormal nerve conduction velocities
* Ability to cooperate for clinical evaluation and repeat nerve conduction studies
* Willingness of sexually active subjects to practice a reliable method of contraception during the study

Exclusion Criteria:

* Active viral infection based on clinical observations or serological evidence of HIV, or Hepatitis B or C infection, herpesvirus or adenovirus
* Ongoing immunosuppressive therapy or immunosuppressive therapy within 6 months of starting the trial (e.g., corticosteroids, cyclosporine, tacrolimus, methotrexate, cyclophosphamide, intravenous immunoglobulin)
* Persistent leukopenia or leukocytosis (WBC ≤ 3.5 K/µL or ≥ 20.0 K/µL) or an absolute neutrophil count < 1.5K/µL
* Subjects with AAV1 binding antibody titers ≥ 1:50 as determined by ELISA immunoassay
* Subjects with circulating anti-NT-3 titers ≥ 1:50 as determined by ELISA immunoassay
* Treat with any investigational medication within 30 days before the infusion of study drug
* Abnormal laboratory values considered clinically significant (GGT > 3XULN, bilirubin ≥ 3.0 mg/dL, creatinine ≥ 1.8 mg/dL, Hgb < 8 or > 18 g/Dl; WBC > 15,000 per cmm)
* Any medical condition or extenuating circumstance that, in the opinion of the investigator, might compromise the subject's ability to comply with the protocol required testing or procedures or compromise the subject's wellbeing, safety, or clinical interpretability
* Ankle contractures or surgeries preventing proper muscle strength testing
* Pregnancy or lactation (females subjects will be tested for pregnancy)
* Limb surgery in the past six months
* Severe infection (e.g. pneumonia, pyelonephritis, or meningitis) within 4 weeks before gene transfer visit (enrollment may be postponed)
* Anyone unwilling to disclose study participation with primary care physician and other medical providers.
* Concomitant illness or requirement for chronic drug treatment that in the opinion of the PI creates unnecessary risks for gene transfer

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2027-04 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Safety based on number of participants with adverse events. | 2 years
  AEs will be monitored and scored for severity and relatedness to the study article.

SECONDARY OUTCOMES:
Efficacy - the ability to halt the decline in functional and sensory abilities | Screening, Day 90, 6 months, 1yr, 18 months, 2 yrs
  CMT Pediatric Scale. Efficacy will be defined as the ability to halt the decline in functional and sensory abilities as measured by the CMTPedS at 2 years post gene transfer. This 11 item scale, developed by the Inherited Neuropathies Consortium, underwent validation testing in patients aged 3-20 years with CMT and generates a linear score of disability.
Physical Therapy Assessments The 100 Meter Timed Test (100m) | Screening, Day 90, 6 months, 1yr, 18 months, 2 yrs
  The 100 Meter Timed Test will be an exploratory outcome for this study.
Electrophysiological testing | Screening, Day 90, 6 months, 1yr, 18 months, 2 yrs
  Measurement of ulnar sensory nerve amplitude and compound muscle action potential (CMAP); amplitude of the ulnar nerve (recorded from the abductor digiti minimi muscle) and the peroneal nerve (recorded from the tibialis anterior muscle) and sensory and motor conduction velocities.
Sensory testing using semi-quantitative Rydel Seiffer tuning fork, Semmes-Weinstein Monofilaments and Neurotips | Screening, Day 90, 6 months, 1yr, 18 months, 2 yrs
  Perceptions of touch pressure, pricking pain and vibration will be graded on the index finger and the great toe as normal (0), decreased (1), or absent (2). In addition, the level of discrimination change for sensory modalities will be recorded in the dominant upper and lower limbs as normal (0), diminished or absent in fingers or toes (1), between fingers/toes and wrist or ankle (2), between wrist/ankle and mid-forearm or mid-calf level (3), between mid-forearm/mid-calf and elbow or knee (4) and above the level of elbow or knee (5).
Visual analog scale (VAS) | Screening, Day 90, 6 months, 1yr, 18 months, 2 yrs
  The visual analog scale (VAS) of pain intensity consists of a line, most often 100 mm long, with 2 descriptors representing extremes of pain intensity (e.g., no pain and extreme pain) at each end. Patients rate their pain intensity by making a mark somewhere on the line that represents their pain intensity and the VAS is scored by measuring the distance from the "no pain" end of the line.
Short Form Health Survey (SF-36) | Screening, Day 90, 6 months, 1yr, 18 months, 2 yrs
  The Short Form Health Survey (SF-36) will be used as a quality of life document to monitor and compare disease burden pre and post-treatment. The SF-36 is a multi-purpose, short-form health survey with only 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index.
NT-3 levels | Screening, Day 7-2 yrs
  Circulating NT-3 levels will be measured by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Zarife Sahenk, MD., PhD., Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States